CLINICAL TRIAL: NCT03046290
Title: Pudendal Block Versus Penian Block For Circumcision In Children: A Double Blind Randomised Controlled Trial
Brief Title: Pudendal Block Versus Penian Block For Circumcision In Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, JOHN NICOLARDOT, MD, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B406201630517; U1111-1191-4760 (Other: WHO UTN)
Record Dates: First submitted 2017-01-10; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Regional Anesthesia; Postoperative Pain; Circumcision
MeSH Terms: conditions — Pain, Postoperative | interventions — Circumcision, Male; Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pudendal Block (Active Comparator): The anesthesia is produced by blocking the pudendal nerves near the ischial spine of the pelvis.Local anesthetic (mixed of ropivacaine and lidocaine) is injected into the pudendal canal where the pudendal nerve is located.
  Interventions: Procedure: circumcision; Drug: Lidocaine; Drug: Ropivacaine
- Penian Block (Active Comparator): The anesthesia is produced by blocking the dorsal penile nerves. Local anesthetic (mixed of ropivacaine and lidocaine)is injected under the pubis symphysis just below the Buck fascia where the nerve is located.
  Interventions: Procedure: circumcision; Drug: Lidocaine; Drug: Ropivacaine

INTERVENTIONS:
Procedure: circumcision
Drug: Lidocaine
Drug: Ropivacaine

SUMMARY:
The authors study the efficacy of the pudendal versus penile block for the relief of postoperative pain in children receiving ambulatory circumcision.

In this prospective, double-blind, randomized, parallel-arm trial, 60 children recruited during the anesthesia consultation will be allocated a general anesthesia with a pudendal block (PUD group) or a penile block (PEN group).

Each block will be made with equal parts lidocaine 1% and ropivacaine 0.75% (0.3 ml/kg).

ELIGIBILITY:
Inclusion Criteria:

* circumcision in day surgery hospital

Exclusion Criteria:

* allergy to amino-amide local anesthetics
* parental consent not received
* infection at injection site

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | pain score at 0 hours postoperatively
  using the FLACC (Face Leg Activity Cry Consolability) Scale

SECONDARY OUTCOMES:
Degree of satisfaction of the patient or his/her parents and the surgeon assessed by telephone interview | Day 5 after the procedure
  telephone interview

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme, Bruxelles Capitale, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naja Z, Al-Tannir MA, Faysal W, Daoud N, Ziade F, El-Rajab M. A comparison of pudendal block vs dorsal penile nerve block for circumcision in children: a randomised controlled trial. Anaesthesia. 2011 Sep;66(9):802-7. doi: 10.1111/j.1365-2044.2011.06753.x. Epub 2011 Jul 25. PMID 21790518
- [Background] Faraoni D, Gilbeau A, Lingier P, Barvais L, Engelman E, Hennart D. Does ultrasound guidance improve the efficacy of dorsal penile nerve block in children? Paediatr Anaesth. 2010 Oct;20(10):931-6. doi: 10.1111/j.1460-9592.2010.03405.x. PMID 20849498
- [Background] O'Sullivan MJ, Mislovic B, Alexander E. Dorsal penile nerve block for male pediatric circumcision--randomized comparison of ultrasound-guided vs anatomical landmark technique. Paediatr Anaesth. 2011 Dec;21(12):1214-8. doi: 10.1111/j.1460-9592.2011.03722.x. PMID 22023417